CLINICAL TRIAL: NCT04888130
Title: Investigation of an Outbreak Situation of Cutaneous Leishmaniasis Among Military Personnel in French Guiana (CEFELEISH)
Acronym: CEFELEISH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Centre Médical Inter-Armées (CMIA) de Cayenne, French Guiana (Unknown); Centre Médical Inter-Armées (CMIA) de Kourou, French Guiana (Unknown); Direction Interarmées du Service de Santé des Armées (DIASS) de Cayenne, French Guiana (Unknown); Centre National de Référence des Leishmanioses, CHU de Montpellier, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: CEFELEISH
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Leishmaniasis, Cutaneous; Risk Factors; Phylogeny; Military Personnel; Prevalence; French Guiana; Outbreak
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Phylogeny; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: This study comes following an outbreak signal that occurred in May 2020, after the detection of numerous cases of cutaneous leishmaniasis in military personnel probably contaminated during a training course (Training Center in the Equatorial Forest, CEFE) in the town of Regina. To date, around 40 cases have been detected.
  Interventions: Genetic: Phylogenetic Analysis; Other: Data collection
- Controls: A case-control study can therefore be carried out using a questionnaire offered to all course participants over the 1st semester of 2020. The controls will then be participants who have not been infected. A comparison can also be made between the military personnel present in French Guiana during the first half of 2020 and having carried out missions in the forest, by opposing the participants and non-participants of the CEFE.
  Interventions: Other: Data collection

INTERVENTIONS:
Genetic: Phylogenetic Analysis — The phylogenetic analysis is carried out on a sample already taken in routine care (smear, culture on biopsy or PCR on swab).
  Groups: Cases
Other: Data collection — Data will be collected using a standardized digital questionnaire, including clinical and microbiological features, treatments received details and training conditions and. Data will then be compared between patients with therapeutic success or failure.

SUMMARY:
Clinical, epidemiological, therapeutic and microbiological investigation of an outbreak of cutaneous Leishmaniasis that occurred among military personnel in French Guiana in 2020.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is endemic in French Guiana and represents 200 to 300 cases per year. Transmission occurs after a sandfly bite, mainly during the rainy season and over almost all of French Guiana. The incidence is, however, greater in forest areas, especially in recently cleared areas. Nevertheless, transmission remains continuous and outbreaks remain rare and little investigated. This study comes following an outbreak signal that occurred in May 2020, after the detection of numerous cases of cutaneous leishmaniasis in military personnel probably contaminated during a training course (Training Center in the Equatorial Forest, CEFE) in the town of Regina. To date, around 40 cases have been detected. This outbreak raises several scientific questions, on the microbiological, clinical and epidemiological level.

From a microbiological point of view, it is not certain whether the occurrence of a large number of cases in a given group over a short period can be attributed to a single leishmania clone or only reflect exposure to a large number of infected sandflies. An L. braziliensis outbreak has been described in naturalists on mission in the Saul region, but it is possible that several species are detected in a larger outbreak. The description of the activities at the origin of the contamination can influence the offending species insofar as the different sandfly species do not use the same reservoirs, are not found in the same ecosystems and do not carry the same species of leishmanias.

Clinically, in the case that many patients are infected after the bite of similar sandflies and under similar conditions, similar clinical manifestations could be expected. It would be interesting to look for variations in terms of the type, number, localization, severity of lesions, and especially of response to treatment, which would reflect the role of factors linked to the host and its immune response. A phylogenetic study would make it possible to compare the strains isolated during this outbreak with other Guyanese isolates from the 2020 rainy season in order to search for a genetic cluster. A comparison can also be made between the strains of the outbreak in order to find a correlation with the clinical severity of certain patients or resistance to first-line treatment (Pentacarinat).

Epidemiologically, the outbreak occurred at a training site already used in previous years, but without such numerous cases being reported. This site sits on 700 hectares of primary forest and has not recently undergone additional development or deforestation. The course of activities and the type of training carried out by the military has not changed this year. A change in environmental conditions and exposure to sandflies therefore does not seem to explain this increase in cases. A capture of sandflies, delayed in relation to the period of contamination, would not allow the question of environmental change to be answered.

On the other hand, looking for behavioral risk factors (clothing, night shower, role played in exercises, type of hammock used, etc.) could provide explanations for the occurrence of infections in some trainees and not in their classmates. A case-control study can therefore be carried out using a questionnaire offered to all course participants over the 1st semester of 2020. The controls will then be participants who have not been infected. A comparison can also be made between the military personnel present in French Guiana during the first half of 2020 and having carried out missions in the forest, by opposing the participants and non-participants of the CEFE, in order to determine whether this course represented an independent risk factor for leishmaniasis. This result would reflect a higher exposure than conventional operations against gold mining, for example.

Investigation of this outbreak would make it possible to take corrective actions in terms of prevention and public health. It would provide a better understanding of the pathophysiological mechanism of contamination (clonal or not) and the consequences in terms of infecting species, clinical severity and expected therapeutic response in the circumstances of grouped cases of cutaneous leishmaniasis.

Retrospective cohort study for the clinical and microbiological part (grouped cases of an outbreak) Case-control section with questionnaires assessing exposure to sandflies National multicenter sample Category 3 Non-Interventional Human Person Research (RIPH 3)

ELIGIBILITY:
* Inclusion criteria

  * for cases :
* Confirmed cutaneous leishmaniasis (compatible clinical lesion + a positive microbiological test or cure after probabilistic anti-leishmania treatment) in a military personnel who participated in the CEFE training

  *for controls :
* Absence of a suspicious lesion of leishmaniasis in a military personnel who participated in training at CEFE

NB: All concerned are adults.

* Non inclusion criteria

  *for cases :
* Confirmed cutaneous leishmaniasis not having been contracted after a training at CEFE
* Unconfirmed cutaneous leishmaniasis
* Opposition to the use of their data and / or the completion of the questionnaire
* Refusal of participation

  *for controls :
* Opposition to the taking of the questionnaire
* Refusal of participation training
* Exclusion criteria Withdrawal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study comes following an outbreak signal that occurred in May 2020, after the detection of numerous cases of cutaneous leishmaniasis in military personnel probably contaminated during a training course (Training Center in the Equatorial Forest, CEFE) in the town of Regina. To date, around 40 cases have been detected.
  A case-control study can therefore be carried out using a questionnaire offered to all course participants over the 1st semester of 2020. The controls will then be participants who have not been infected. A comparison can also be made between the military personnel present in French Guiana during the first half of 2020 and having carried out missions in the forest, by opposing the participants and non-participants of the CEFE.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Severity of leishmaniasis | 5 months
  • For the cohort study part: Primary endpoint: severity of leishmaniasis (clinical presentation, cure after Pentacarinat) Associations will be sought between this main criterion and the phylogeny of the strains and the patient's intrinsic risk factors.

OTHER OUTCOMES:
Frequency of responses collected during questionnaire | 5 months
  • For the case-control part: Primary endpoint: comparison of the frequency of responses collected during the questionnaire between cases and witnesses

CONTACTS AND LOCATIONS:
Overall Officials: DEMAR PIERRE Magalie, PhD, Study Director — Centre Hospitalier de Cayenne
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

REFERENCES:
- [Background] Loiseau R, Nabet C, Simon S, Ginouves M, Brousse P, Blanchet D, Demar M, Couppie P, Blaizot R. American cutaneous leishmaniasis in French Guiana: an epidemiological update and study of environmental risk factors. Int J Dermatol. 2019 Nov;58(11):1323-1328. doi: 10.1111/ijd.14625. Epub 2019 Sep 16. PMID 31524286
- [Background] Simon S, Nacher M, Carme B, Basurko C, Roger A, Adenis A, Ginouves M, Demar M, Couppie P. Cutaneous leishmaniasis in French Guiana: revising epidemiology with PCR-RFLP. Trop Med Health. 2017 Feb 28;45:5. doi: 10.1186/s41182-017-0045-x. eCollection 2017. PMID 28265182
- [Background] Martin-Blondel G, Iriart X, El Baidouri F, Simon S, Mills D, Demar M, Pistone T, Le Taillandier T, Malvy D, Gangneux JP, Couppie P, Munckhof W, Marchou B, Ravel C, Berry A. Outbreak of Leishmania braziliensis Cutaneous Leishmaniasis, Saul, French Guiana. Emerg Infect Dis. 2015 May;21(5):892-4. doi: 10.3201/eid2105.141181. No abstract available. PMID 25897573